CLINICAL TRIAL: NCT01256255
Title: INFLUENZA VIRUS INFECTIONS IN TRANSPLANT RECIPIENTS: A MULTICENTER REGISTRY
Brief Title: Influenza Virus - A Multicenter Registry
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: UOA-FLU-2010-11
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Influenza Infection in Transplant Patients
Keywords: transplant; influenza infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and nasal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- influenza infection: Patients with the diagnosis of influenza infection by standard laboratory technique

SUMMARY:
The investigators purpose is to prospectively characterize influenza infections over a 3 year period in transplant patients using a registry system. The investigators plan to generate robust data on clinical features of upper and lower respiratory disease, antiviral therapy and its effects on disease outcome, as well as quantitative virologic data on shedding and antiviral resistance. The investigators also will study the long term sequelae of influenza infections and look at development of rejection.

DETAILED DESCRIPTION:
This study will be a prospective, multi-center study conducted at investigator sites who comprise the Influenza in Transplant collaborative study group. This includes over 30 centers from across North America and Europe. The co-ordinating center will be the University of Alberta. We will aim to enrol 300 patients in the registry over a 3 year period.

The following information will be gathered:

1. Clinical Information

   * Baseline demographic information about the transplant (including immunosuppression, graft function)
   * Comorbidities such as diabetes, obesity, chronic lung disease
   * Symptoms of infection, radiologic features of infections
   * Antiviral use
   * History of vaccination
   * Outcomes such as hospitalization, ICU admission, mechanical ventilation, death
   * Long term outcomes: allograft function, chronic respiratory disease
   * Laboratory parameters including lymphocyte count, immunoglobulin levels, renal function
   * Adverse events - all serious adverse events occurring during the study (till day 180) will be reported. These include: a) hospitalization; b) congenital deformity; c) death; d) disability; and e) other adverse events the investigator considers serious. Pregnancy during the follow-up period will also be reported.
2. Virology

   * Method of diagnosis (DFA, viral culture, PCR)
   * Subtype of influenza virus (ie HxNx)
   * Viral Shedding by serial NP swabs at day 0 (diagnosis), 3, 6, 11, 18, 28 (weekly thereafter if shedding persists)
   * Quantitative PCR of NP swabs (centrally at University of Alberta)
   * Antiviral resistance testing at first and last positive swabs
3. Immunology - Serum collection at disease onset and 4-6 weeks afterwards for

   * Serology against circulating influenza viruses
   * Production of HLA alloantibodies

Significance:

Despite the recognized importance of influenza in transplant patients, there is actually very limited prospective data. This registry will represent the largest prospective data collection on influenza in transplant patients and will provide invaluable data on the clinical presentations, antiviral efficacy and other parameters related to influenza.

ELIGIBILITY:
Inclusion Criteria:

* Solid organ transplant recipients on at least one immunosuppressive medication
* Hematopoietic stem cell transplant recipients - allogeneic or autologous
* Pediatric or Adult
* Diagnosis of influenza infection by standard laboratory technique

Exclusion Criteria:

not able to comply with the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Solid organ transplant recipients on at least one immunosuppressive medication and Hematopoietic stem cell transplant recipients (allogeneic or autologous) with the diagnosis of influenza infection by standard laboratory technique
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2010-11; Primary Completion 2013-08-31 (Actual); Study Completion 2014-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] L'Huillier AG, Ferreira VH, Hirzel C, Cordero E, Limaye AP, Reid G, Englund J, Blumberg E, Kumar D, Humar A. Cytokine Profiles and Severity of Influenza Infection in Transplant Recipients. J Infect Dis. 2019 Jan 29;219(4):535-539. doi: 10.1093/infdis/jiy535. PMID 30192949